CLINICAL TRIAL: NCT05226494
Title: A Phase 1 Trial to Evaluate the Safety and Tolerability of Fb-PMT in Patients With Recurrent Glioblastoma
Brief Title: Safety and Tolerability of Fb-PMT in Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NanoPharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NP-100-101
Record Dates: First submitted 2021-12-03; First posted 2022-02-07 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Glioma, Malignant
Keywords: Glioblastoma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Intervention Model Description: 3+3 Dose Escalation with option for cohort expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (fb-PMT) (Experimental): Daily subcutaneous injection of fb-PMT in four escalating cohorts to determine maximum tolerated dose, followed by treatment of up to 10 additional patients at maximum tolerated dose.
  Interventions: Drug: fb-PMT

INTERVENTIONS:
Drug: fb-PMT — Daily dosing based on patient weight
  Other Names: NP-100; NP751

SUMMARY:
Glioblastoma is a highly aggressive and fatal form of primary malignant brain tumor with limited treatment options. fb-PMT affects a large group of cancer cell signaling pathways and thus may be effective in heterogeneous, treatment-resistant tumors such as Glioblastoma. fb-PMT also is actively transported across the blood-brain barrier into the brain. This study is being conducted to determine the dose level for further clinical development of fb-PMT to treat recurrent Glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven intracranial glioblastoma, with first or second recurrence
* On stable or decreasing dose of steroids, if taken prior to screening
* Baseline MRI (with and without contrast) completed with 5 days of starting fb-PMT
* Prior completion of and recovery from the effects of standard of care for glioblastoma management with surgery/biopsy and radiotherapy
* Confirmation of true progressive disease for patients previously treated with interstitial brachytherapy or stereotactic radio surgery
* Life expectancy of more than three months
* Karnofsky Performance Status of ≥ 70
* Hypertension must be well controlled (≤ 95th percentile) on stable doses of medication
* Adequate bone marrow and organ function, confirmed by laboratory testing at screening
* Patient or caregiver must be able to store drug under refrigerated conditions, prepare and administer daily subcutaneous injections on a set schedule, and record information in a daily treatment diary
* Women of childbearing potential must agree to ongoing pregnancy testing and to use medically acceptable contraception for the duration of the study and for 2 months after their last dose of study drug
* Males must agree to use medically acceptable contraception and refrain from donating sperm for the duration of the study and for 2 months after their last dose of study drug

Exclusion Criteria:

* Significant medical illness that is uncontrolled, may obscure toxicity, may dangerously alter drug metabolism, or may compromise ability for study participation
* History of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off all therapy for that disease for at least 3 months prior to first dose of study drug
* Use of bevacizumab or any other experimental drug or therapy within 28 days of study treatment
* Prior therapy with fb-PMT or related drugs
* Currently pregnant or breastfeeding
* Active infection or serious intercurrent medical illness
* Surgery of any type within the preceding 28 days that has not fully healed
* A serious or non-healing wound, ulcer, or bone fracture
* A known bleeding diathesis or coagulopathy, or a history of bleeding diathesis within 28 days of study treatment
* A known thrombophilic condition (i.e., protein S, protein C, or antithrombin III deficiency, Factor V Leiden, Factor II G20210A mutation, homocysteinemia or antiphospholipid antibody syndrome). Testing is not required in patients without thrombophilic history.
* Evidence of new central nervous system hemorrhage on baseline MRI obtained within 14 days prior to study enrollment
* Clinically significant cardiovascular event such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening.
* New York Heart Association classification of heart disease greater than Class 2
* QTc interval > 450 msec in males or > 470 msec in females at screening
* Use of concomitant medications that prolong the QT/QTc interval or risk inducing Torsades de Pointes
* Use of any concomitant OATP1B1, OATP1B3, or BSEP inhibitors within 14 days or five half-lives (whichever is longer) before starting study drug treatment
* Abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within 6 months prior to study enrollment
* A significant vascular disease (e.g., aortic aneurysm requiring surgical repair, deep venous or arterial thrombosis) within the last 6 months prior to study enrollment
* History of stroke, myocardial infarction, transient ischemic attack (TIA), severe or unstable angina, peripheral vascular disease, or grade II or greater congestive heart failure within the past 6 months
* History of Torsades de Pointes or risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 15 months
  Determined by the number of Treatment-Emergent Adverse Events, including Dose-Limiting Toxicities per patient.
Incidence of Dose Limiting Toxicities [Safety and Tolerability] | 28 Days
  Number of participants with a dose-limiting toxicity during the first cycle (28 days) of treatment at their highest dose level administered.

SECONDARY OUTCOMES:
Establishment of Recommended Phase 2 Dose | 28 Days
  Maximum Tolerated Dose, as determined by Dose-Limiting Toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Blondin, MD, Principal Investigator — Yale University
Locations (1):
- Smilow Cancer Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No